CLINICAL TRIAL: NCT05433506
Title: A Phase 1, Two-Part Study to Assess the Safety and Pharmacokinetics of Tablet and Capsule Formulations of HU6 in Obese Subjects.
Brief Title: Safety and Pharmacokinetics of HU6
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RIV-HU6-103
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Part 1 is an open-label, randomized, Latin-square 2x2 crossover study. Part 2 is an open-label study of up to 4 single, ascending dose levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment: HU6 Tablet (Experimental)
  Interventions: Drug: HU6 Tablet
- Active Treatment: HU6 Capsule (Experimental)
  Interventions: Drug: HU6 Capsule

INTERVENTIONS:
Drug: HU6 Tablet — Six subjects will receive a tablet formulation.
  Arms: Active Treatment: HU6 Tablet
Drug: HU6 Capsule — Six subjects will receive the capsule formulation
  Arms: Active Treatment: HU6 Capsule

SUMMARY:
Part 1 is an open-label, randomized, Latin-square 2x2 crossover study. Twelve subjects will be randomized (1:1) to treatment sequence to determine the order in which they will receive the tablet or capsule formulation in Period 1 and Period 2.

Part 2 is an open-label study of up to 4 single, ascending dose levels of HU6 administered as the tablet formulation. Eight subjects will be enrolled to participate in all of the ascending study periods.

DETAILED DESCRIPTION:
Part 1 is an open-label, randomized, Latin-square 2x2 crossover study. Twelve subjects will be randomized (1:1) to treatment sequence to determine the order in which they will receive the tablet or capsule formulation in Period 1 and Period 2. There will be a minimum 10 day washout period between dosing in Period 1 and Period 2.

Part 2 is an open-label study of up to 4 single, ascending dose levels of HU6 administered as the tablet formulation. Eight subjects will be enrolled to participate in all of the ascending study periods. There will be a minimum 14-day washout period between dosing in each study period. The washout is longer in Part 2 to allow time for pharmacokinetic analyses and data review between study periods.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female between 18 and 55 years of age, inclusive, at time of informed consent.

  1. Female subjects of childbearing potential must be non-lactating, not pregnant as confirmed by a negative urine serum pregnancy test at Screening and admission to CRU, and using, and agree to continue using, an effective method of contraception for at least 4 weeks or barrier method for 2 weeks prior to first study drug administration until 30 days after the last dose of study drug.
  2. Female subjects of non-childbearing potential must be surgically sterile (e.g., hysterectomy, bilateral tubal ligation, oophorectomy) or post-menopausal (no menses for >1 year with follicle stimulating hormone (FSH) >40 U/L at Screening).
  3. Female subjects of childbearing potential must not donate ova during the study and for at least 30 days after the last dose of study drug.
  4. Male subjects who have not had a vasectomy and/or subjects who have had a vasectomy but have not had 2 post surgery negative tests for sperm must agree to use an acceptable method of contraception from time of first dose of study drug until 30 days after the last dose of the study drug, and to not donate sperm during the study and for at least 30 days after the last dose of study drug.

     2. BMI between 28.0 and 45.0 kg/m2, inclusive. 3. Healthy per investigator judgment as documented by medical history, physical examination, vital sign assessments, 12-lead ECG, clinical laboratory assessments, and general observations. Note that Screening, abnormalities or findings outside the normal ranges for any clinical assessments that are considered clinically significant by the Investigator (clinical laboratory tests, ECG, vital signs) may be repeated once at the discretion of the Investigator(s), and results that continue to be outside the normal ranges must be judged by the investigator to be not clinically significant and acceptable for study participation.

     4. Able to understand the procedures and requirements of the study and provide written informed consent and authorization for protected health information disclosure.

     5. Willing and able to comply with the requirements of the study protocol.

     Exclusion Criteria:
* Subjects presenting with any of the following will not qualify for entry into the study:

  1. Current or past clinically significant history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, as determined by the investigator in consultation with the medical monitor, which may impact safety. History of cancer (except treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to Screening.
  2. Any surgical or medical condition or history that, in the opinion of the investigator in consultation with the medical monitor, may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to, gastric bypass surgery or significant small bowel resections.
  3. Contraindication to study drug or its excipients and/or history of allergic or anaphylactic reactions or clinically significant allergic reaction.
  4. Resting heart rate <45 or >100 bpm, systolic blood pressure <90 or >160 mm Hg, or diastolic blood pressure <50 or >110 mmHg.
  5. On screening ECG and by history:

     1. A marked baseline prolongation of QT/QTcF interval (e.g., repeated demonstration of a QTcF interval >450 msec for males and >470 msec for females).
     2. A history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) or a family history (immediate family member or grandparent < 60 years of age) of sudden cardiac death of unknown origin.
  6. Use of any prescription medication or over-the counter medications (including multivitamins, herbal-containing preparations and products with cannabidiol [CBD]) within 14 days prior to admission to CRU.

     Exceptions:
     1. Hormonal contraceptives and hormone replacement therapies (oral, injectable, transdermal, or implanted) are permitted.
     2. Topical medication for skin disorders may be added at the discretion of the PI in consultation with the Medical Monitor, if it is determined there is no significant systemic absorption of the medication which may impact other exclusions of medications noted above.
     3. Acetaminophen may be taken during screening and as needed to treat an AE during the study, but subjects should not receive acetaminophen within 24 hours of admission to the CRU.
     4. Ibuprofen (or other nonsterioidal anti-inflammatory drug [NSAID]) is prohibited within 7 days prior to admission to the CRU.

     c)
  7. Consumption of any food or drink/beverage containing grapefruit or grapefruit juice, apple or orange juice, pomelo juice, star fruit, Seville or Moro (blood) orange products within 7 days before admission to CRU. Vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard), food containing poppy seeds (e.g., muffins, bagels, and cakes) must not be consumed within 24 hours before admission to CRU.
  8. History of significant drug abuse (i.e, cocaine, phencyclidine, opioid derivatives including heroin, and amphetamine derivatives)within one year prior to Screening or frequent use of soft drugs (such as marijuana) within 1 month prior to the Screening visit, or hard drugs (such as cocaine, phencyclidine, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening. Marijuana use (and other tetrahydrocannabinol [THC] containing products) is prohibited within 7 days prior to Screening and throughout the study. .
  9. History of regular alcohol consumption exceeding 14 drinks/week [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months of Screening.
  10. Positive urine drug screen for drugs of abuse or positive phosphatidylethanol (PEth) blood test result >200 ng/mL based on PEth 16.0/18.1 (POPEth) at Screening or on admission to the CRU. In instances of an exclusionary PEth value, consideration for enrollment/study continuation can be provided if the principal investigator and medical monitor agree the subject's history is not consistent with alcohol abusePositive urine drug or urine alcohol test at Screening or on admission to CRU.
  11. Current nicotine use or vaping regularly more than 5 cigarettes or the equivalent per week. Use of nicotine patches for smoking cessation is not permitted within 7 days of dosing.
  12. Positive test results of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV1/2) antibody.
  13. Diabetes, reflected by a fasting plasma glucose level of ≥126 mg/dL andor a reflex hemoglobin A1c (HbA1c) ≥6.5%.
  14. Neutropenia, defined as absolute neutrophil count ≤1000/µL.
  15. Participation in another clinical trial at the time of screening or exposure to any investigational agent, including topical agents, within 30 days or 5 half-lives prior to admission to CRU, whichever is longer.
  16. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
  17. Having a condition that the investigator believes would interfere with his/her ability to provide written informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk. Subjects with a history of hypo- or hyperthyroidism, peripheral neuropathy, malignant hyperthermia, cataracts or chronic recurrent rash that is considered clinically significant by the investigator are excluded.
  18. Familial (mother/father/sibling) and/or personal history of retinal detachment any time in the past.
  19. Evidence of the following on screening ophthalmologic examination:

      1. Peripheral retinal pathology requiring treatment, retinal tears, or lattice that require treatment.
      2. Diabetic retinopathy with macula exudates or macula edema as shown by optical coherence tomography and examination.
      3. Any active macular disease that affects the vision, including macula pucker (epiretinal membrane) and macular degeneration.
      4. Visually significant cataract as determined by ophthalmologist.
      5. Any previous intravitreal injection of anti-VEGF agents for macular degeneration.
      6. History of prior vitrectomy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Assess the dose relationship of PK Parameter Cmax | 150 days
  Following completion of each cohort, bioanalytical and the PK parameter Cmax will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Ferrer, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided